CLINICAL TRIAL: NCT03173846
Title: Multiregional rtfMRI Neurofeedback for the Prevention of Alzheimer's Disease
Brief Title: Multiregional rtfMRI Neurofeedback for the Prevention of Alzheimer's Disease (NPAD)
Acronym: NPAD
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ALFA-NPAD/BBRC2016
Record Dates: First submitted 2017-05-29; First posted 2017-06-02 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease
Keywords: neurofeedback; episodic memory; real-time functional MRI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult children of AD patients

SUMMARY:
This study aims to predict cognitive decline using a performance endophenotype of neuro-feedback based on functional magnetic resonance imaging in real time in a population at risk for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
In this research project, a longitudinal study in a healthy population that is under increased risk of developing AD will be performed. It is anticipated that some of the participating subjects will develop episodic memory decline within this longitudinal follow-up. The memory binding Test (MBT) and/or the Free and Cued Selective Reminding Test (FCSRT), the most accurate and reliable available episodic memory tests, are going to be performed by the subjects at multiple longitudinal data collection points. The project proposes to develop a real-time functional magnetic resonance imaging (rtfMRI) task, and to test whether the subjects' performance on the task can predict the apparition of cognitive decline. The impact of other relevant biomarkers by adding them to the model: age, gender, number of APOE-e4 alleles, cognitive scores, cerebrospinal fluid (CSF) biomarkers, amyloid Positron Emission Tomography (PET), lifestyle habits and clinical background will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (aged 45-75) that have participated in the study 45-65/FPM2012.
* Persons that accept the study's test and procedures that are as follows: magnetic resonance imaging and neuropsychological tests.
* Signature of the study's informed consent form, accepting to not receive information with regards to any research results that are not clinically relevant.

Exclusion Criteria:

* Any contraindication to MRI (e.g. pacemaker, claustrophobia, etc.)
* Any condition that according to the investigator's judgement could interfere with the proper execution of the study's procedures and/or its follow-up.

Ages: 45 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participating subjects are healthy adults (aged 45-75 at inclusion) already recruited within the ALFA study (http://clinicaltrials.gov/ct2/show/NCT01835717; Estudi 45-65 FPM/2012).
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cognition | 12 months
  Predictive value of neurofeedback performance

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No